CLINICAL TRIAL: NCT02805764
Title: Changes in Upper Airway Anatomy, Quality of Life Measures, and Polysomnographic Parameters Using A Functional Dental Appliance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No suitable candidates
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Steven Y. Park, Attending Surgeon / Assistant Professor - Otorhinolaryngology, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-4845
Record Dates: First submitted 2016-05-31; First posted 2016-06-20 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea; Malocclusion
Keywords: obstructive sleep apnea; malocclusion; polysomnography; quality of life
MeSH Terms: conditions — Sleep Apnea, Obstructive; Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Homeoblock functional dental appliance (Experimental): Removable functional dental appliance to be used at during sleep for one year.
  Interventions: Device: Homeoblock

INTERVENTIONS:
Device: Homeoblock — A removable, functional dental appliance to be worn nightly for 1 year Pending 510(k) clearance for the use of reducing snoring and mild to moderate obstructive sleep apnea in adults. A class II medical device.

SUMMARY:
A prospective study measuring changes in upper airway anatomy, quality of life measures, and polysomnographic parameters using a functional dental appliance (Homeoblock)

DETAILED DESCRIPTION:
Although rising levels of obesity heavily influences the increasing rates of obstructive sleep apnea (OSA), detailed analysis of more basic etiology suggests a possible craniofacial origin. Specifically, modern humans' facial structures a slowly shrinking, which can narrow the upper airway. This is evidenced by the fact that rates of malocclusion and impacted (or non-existent) wisdom teeth are increasing in modern, Westernized countries.

Obstructive sleep apnea is a commonly seen condition characterized by multiple episodes of obstructed breathing during sleep, with intermittent hypoxia. Untreated OSA is associated with significantly higher rates of high blood pressure, diabetes, heart disease, heart attack, stroke, sudden death, and car accidents. The gold standard treatment for OSA is continuous positive airway pressure (CPAP), but compliance is poor. Initially, out of 100 patients, 20 will refuse CPAP. After one year 50% of the 80 remaining patients will be using CPAP, but only 50% will be using it effectively, leaving only 20 patients who are using CPAP effectively. (personal communication, Stepnowski).

An alternative option in people with mild to moderate OSA is a mandibular advancement device, which functions by pulling the genioglossus muscle forward. Long-term use of CPAP and mandibular advancement devices have been shown to aggravate malocclusion. Numerous surgical options are available for select patients, but only as a last resort.

In children, one uncommonly used, but effective form of treating OSA is by application of a palatal expander by an orthodontist. In theory, this option is effective due to the fact the palatal suture line is not completely fused in children. The general consensus in dentistry is that adults have fused midline palatal suture line and the hard palate cannot be expanded.

Recent work by numerous investigators suggests that palatal expansion can occur to significant degrees, even in adults. Case reports have been published with the AHI diminishing significantly after therapy. Not only can the hard palate widen, there can also be significant growth of new maxillary bone growth and anterior mandibular bone growth. Jaw development is linked to airway development.

The Homeoblock is once such appliance that is based on principles of epigenetics. Mechanical stimulation by the device is thought to initiate gene transcription within the periodontal ligament, creating dental movement and new bone formation.

Our study aims to determine the efficacy of the Homeoblock in patients with obstructive sleep apnea with regards to changes in polysomnographic parameters, functional quality of life measures, and upper airway anatomy size using low-dose CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Documented AHI > 15 on polysomnography
* Refuses CPAP
* Able to fill our QOL and sleep questionnaires (pre and one year post treatment)
* Willing to undergo CBCT radiologic testing x 2 (pre and 1 year post treatment)

Exclusion Criteria:

* neurologic conditions
* dementia
* central sleep apnea
* heart failure, seizures
* age < 18
* severe nasal congestion
* insufficient teeth
* lack of manual dexterity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-01-02 (Estimated); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Polysomnographic (PSG) parameters, mainly AHI and O2 desaturation measures | Through study completion. Data to be re-collected after one year of therapy for each participant
  Comparison of PSG data between pre-therapy and post-therapy values at one year

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | Comparison of data between pre-therapy and post-therapy values at one year for each participant
  Commonly used validated tool for sleep research
Functional Outcome of Sleep Questionnaire (FOSQ) | Comparison of data between pre-therapy and post-therapy values at one year for each participant
  Commonly used validated tool for sleep research
Nasal obstruction symptom evaluation (NOSE) | Comparison of data between pre-therapy and post-therapy values at one year for each participant
  Commonly used validated tool for otolaryngology research
Upper airway volume changes based on low-dose CT imaging (CBCT) | Comparison of CBCT data between pre-therapy and post-therapy values at one year
  Various upper ariway volume measurements as well as craniofacial landmarks Orthodontists routinely perform periodic CBCT imaging to assess progress. A one year interval is well within standards of care.
BMI | Comparison of data between pre-therapy and post-therapy values at one year

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kushida CA, Efron B, Guilleminault C. A predictive morphometric model for the obstructive sleep apnea syndrome. Ann Intern Med. 1997 Oct 15;127(8 Pt 1):581-7. doi: 10.7326/0003-4819-127-8_part_1-199710150-00001. PMID 9341055
- [Background] Corruccini RS. An epidemiologic transition in dental occlusion in world populations. Am J Orthod. 1984 Nov;86(5):419-26. doi: 10.1016/s0002-9416(84)90035-6. PMID 6594064
- [Background] Chen H, Lowe AA, de Almeida FR, Fleetham JA, Wang B. Three-dimensional computer-assisted study model analysis of long-term oral-appliance wear. Part 2. Side effects of oral appliances in obstructive sleep apnea patients. Am J Orthod Dentofacial Orthop. 2008 Sep;134(3):408-17. doi: 10.1016/j.ajodo.2006.10.031. PMID 18774087
- [Background] Li KK, Riley RW, Guilleminault C. An unreported risk in the use of home nasal continuous positive airway pressure and home nasal ventilation in children: mid-face hypoplasia. Chest. 2000 Mar;117(3):916-8. doi: 10.1378/chest.117.3.916. PMID 10713032
- [Background] Machado-Junior AJ, Zancanella E, Crespo AN. Rapid maxillary expansion and obstructive sleep apnea: A review and meta-analysis. Med Oral Patol Oral Cir Bucal. 2016 Jul 1;21(4):e465-9. doi: 10.4317/medoral.21073. PMID 27031063
- [Background] Singh GD, Callister JD. Effect of a maxillary appliance in an adult with obstructive sleep apnea: a case report. Cranio. 2013 Jul;31(3):171-5. doi: 10.1179/crn.2013.027. PMID 23971157
- [Background] Singh GD, Wendling S, Chandrashekhar R. Midfacial development in adult obstructive sleep apnea. Dent Today. 2011 Jul;30(7):124-7. No abstract available. PMID 21845821
- [Background] Belfor TR, Singh GD. Developing dental arch symmetry using the Homeoblock device. Int J Orthod Milwaukee. 2004 Fall;15(3):27-30. No abstract available. PMID 15553991